CLINICAL TRIAL: NCT05350683
Title: Effect of Remote Ischemic Preconditioning on the Incidence of Contrast Induced Nephropathy in Patients Undergoing EVAR
Acronym: RIPC-EVAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery (Network)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VascularInvestigationNSEACV
Record Dates: First submitted 2022-04-13; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Aortic Aneurysm; Ischemic Preconditioning
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): EVAR patients no ischemic preconditioning
- Preconditioning Group (Active Comparator): EVAR patients with remote ischemic preconditioning
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — In the 12 hours prior to surgery, the principal investigator performed the remote ischemic preconditioning (RIPC) following the protocol: 4 cycles of inflation/deflation of a pneumatic arterial tourniquet on the non-dominant upper extremity. Considering inflated a pressure of 50mmHg above systolic blood pressure for 5 minutes, followed by 5 minutes of deflation. Patients included in the preconditioning group were randomized at a rate of 1:1 consecutively.
  Arms: Preconditioning Group

SUMMARY:
Introduction: Contrast induced nephropathy (CIN) is a major inconvenience in the use of iodinated contrast media (ICM) and it is associated with a significant increase in morbimortality and cost of hospitalization. Remote ischemic preconditioning (RIPC) is a non-invasive and cost-effective tissular protection technique that has proven beneficial in decreasing renal insult in patients receiving intravascular contrast. Aim: The primary outcome of this study is to evaluate the impact of RIPC on the incidence of CIN in patients undergoing endovascular aneurysm repair.Material and Methods: Patients suffering from aortic aneurysm were recruited prior to the administration of iodinated contrast media. Randomization was used to assign patients into the control/RIPC groups. Biochemical parameters determined renal function before and after surgery in immediate (24-72 hours) and at 30 days' follow-up.

DETAILED DESCRIPTION:
2.1. VARIABLES ANALYZED

A randomized prospective study of patients undergoing endovascular treatment for infrarenal abdominal aortic aneurysm, thoracoabdominal aortic aneurysm, descending aortic aneurysm and aneurysms of the aortoiliac sector was designed. These patients were operated at the University Clinical Hospital of Valladolid, in the period between January 2017 and January 2019. The study, which received no financial support from the industry, was performed in agreement with the Declaration of Helsinki and was approved by the institutional review board at each participating site (PI 20-1745, Valladolid East Ethics Committee for Clinical Investigation). In accordance with institutional and local regulatory policies, all patients who underwent procedures within this study signed an informed written consent.

This study only included patients scheduled for elective aortic surgery treated by endovascular repair. On the other hand, exclusion criteria were applied in patients who had peripheral artery disease in the upper limbs, chronic kidney disease grade V on replacement therapy with haemodialysis, patients with cardiac decompensation at the time of the intervention and those who did not tolerate the preparation by ischemic preconditioning in the non-dominant upper limb or who refused to participate in the study.

The variables studied were age and gender, personal history of arterial hypertension, diabetes mellitus, chronic kidney disease and congestive heart failure, levels of estimated glomerular filtrate with the CKD-EPI formula, drugs that may affect renal function such as nephrotoxic medication (metformin, NSAIDs, aminoglycosides, glibenclamide or others) and drugs that can modify renal response to iodinated contrast (n-acetylcystein or sodium bicarbonate) and laboratory values: preoperative serum albumin creatinine, urea, hematocrit and urinary albumin/creatinine ratio in the preoperative period, at 24h and 48h of the administration of iodinated contrast and one month after the administration of iodinated contrast. Volume of iodinated contrast used, intraoperative serum therapy and during admission, type of endograft used, anesthetic technique, intraoperative drugs and in the immediate postoperative period and diuresis in the first 24h was also noted. The impact of preconditioning was measured in terms of absolute and relative creatinine variation in the first 48h according to the definition of contrast nephropathy detailed in section 1.

2.2. NEPHROPROTECTION PROTOCOL

Within 12 hours prior to admission, fluid therapy was administered to all patients in order to prevent the onset of contrast nephropathy. The protocol was applied to all patients regardless of their risk (calculated with the Mehran risk scale) 21, with a regimen of 1ml/kg/hours for 12 hours before surgery. No other nephroprotective drugs such as N-acetylcystin or sodium bicarbonate were used unless the patient required them by prescription of another specialist. Nephrotoxic drugs were removed 24 hours before surgery (NSAIDs, metformin, aminoglycosides and glibenclamide).

2.3. PRECONDITIONING PROTOCOL

In the 12 hours prior to surgery, the principal investigator performed the remote ischemic preconditioning (RIPC) following the protocol: 4 cycles of inflation/deflation of a pneumatic arterial tourniquet on the non-dominant upper extremity. Considering inflated a pressure of 50mmHg above systolic blood pressure for 5 minutes, followed by 5 minutes of deflation. Patients included in the preconditioning group were randomized at a rate of 1:1 consecutively.

2.4. ENDPOINTS

The primary end point of this analysis was to determine 48h and 30-day postoperative CIN (using the above mentioned definition of an absolute increase of >0.5 mg/dl;44μmol/L or a relative increase of >25% of the serum creatinine between 48 - 72 hours after administration of iodinated contrast) in patients with aortic aneurysm who underwent endovascular repair.

Hematocrit levels and urinary albumin:creatinine ratio at 48h and 30-day were also analyzed as secondary endpoints.

2.5. STATISTICAL ANALYSIS

The sample size calculation based on the difference in mean serum creatinine during postoperative period being 0.7 mg/dl between control and RIPC group 19 in a population similar to that of our study. If these assumptions are correct, 37 patients per group would be sufficient to detect a difference of 0,5mg/dl in serum creatinine as defined by the Spanish Society of Nephrology 22. with a power of 80% and a two-sided type 1 error rate of 5% (GRANMO 5.2 statistical software). At the time 18 patients were recruited in each group, standard deviation of the population was 0.7, so a simple size recalculation was mandatory and resulted in 65 patients included in each group of treatment. We estimated 10% loss during follow-up.

Normally distributed continuous variables are summarized with mean and standard deviation and compared using independent group t-tests for continuous variables and ANOVA for numeric variables with repeated values when the data were normally distributed; otherwise, the Mann-Whitney test was used. Continuous variables were tested for normality using the Shapiro-Wilk's test. Categorical variables were expressed as frequencies and percentages and compared by Pearson's chi-square or Fisher's exact test.

For the binary outcomes concerning CIN within 30 days of endovascular aneurysm repair, univariate and multivariate logistic regressions were used. In the multivariate models, patient characteristics, comorbidities, and postoperative complications were used as covariables. Univariate and multivariate logistic regression analyses were performed, and odds ratios (ORs) with 95% confidence intervals (CIs) were reported. Two-sided P values<0.05 were considered statistically significant throughout. All the analyses were performed with the SPSS statistical software package (version 27.0; IBM Corporation, Somers, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective aortic surgery treated by endovascular repair

Exclusion Criteria:

* peripheral artery disease in the upper limbs
* chronic kidney disease grade V on replacement therapy with haemodialysis, - - patients with cardiac decompensation at the time of the interventio
* those who did not tolerate the preparation by ischemic preconditioning in the non-dominant upper limb or who refused to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast induces nephropathy in patients udergoing evar | 48 hours
  serum creatinine
Incidence of contrast induces nephropathy in patients udergoing evar | 30 days
  serum creatinine
Incidence of contrast induces nephropathy in patients udergoing evar | 48 hours
  Estimated glomerular filtrate
Incidence of contrast induces nephropathy in patients udergoing evar | 30 days
  Estimated glomerular filtrate

SECONDARY OUTCOMES:
Other variables | 48 hours
  urinary albumin:creatinine ratio
Other variables | 48 hours
  Hematocrit levels
Other variables | 30 days
  urinary albumin:creatinine ratio
Other variables | 30 days
  Hematocrit levels

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gutierrez, Principal Investigator — Member; Enrique San Norberto, Study Director — Member; Elena Garcia, Study Chair — Member; Liliana Domingos, Study Chair — Member; Cintia Flota, Study Chair — Member; Carlos Vaquero, Study Director — Member
Locations (1):
- Hospital Clínico Universitario, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No